CLINICAL TRIAL: NCT07232290
Title: An Open Label, Randomized, Parallel Controlled, Multicenter Phase IIa Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Flonoltinib Maleate Tablets in the Treatment of Hydroxyurea or Interferon Resistant/Intolerant Polycythemia Vera
Brief Title: Phase IIa Study on Flonoltinib Maleate Tablets in the Treatment of Patients With Polycythemia Vera
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FM-PV-01
Record Dates: First submitted 2025-09-24; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Polycythemia Vera (PV)
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose exploration stage group 1 (Experimental): Flonoltinib 75mg
  Interventions: Drug: Flonoltinib 75mg
- Dose exploration stage group 2 (Experimental): Flonoltinib 100mg
  Interventions: Drug: Flonoltinib 100mg
- Dose exploration stage group 3 (Experimental): Flonoltinib 125mg
  Interventions: Drug: Flonoltinib 125mg
- Extended Phase Dose Group (Experimental): Based on the safety, efficacy, and pharmacokinetic results of the comprehensive dose exploration stage，Flonoltinib xxmg，QD
  Interventions: Drug: Extended Phase Dose Group

INTERVENTIONS:
Drug: Flonoltinib 75mg — Flonoltinib Maleate Tablet 75mg, oral administration, once daily, given on an empty stomach for 8 consecutive weeks of treatment.
  Arms: Dose exploration stage group 1
Drug: Flonoltinib 100mg — Flonoltinib Maleate Tablet 100mg, oral administration, once daily, given on an empty stomach for 8 consecutive weeks of treatment.
  Arms: Dose exploration stage group 2
Drug: Flonoltinib 125mg — Flonoltinib Maleate Tablet 125mg, oral administration, once daily, given on an empty stomach for 8 consecutive weeks of treatment.
  Arms: Dose exploration stage group 3
Drug: Extended Phase Dose Group — Based on the safety, efficacy, and pharmacokinetic results of the comprehensive dose exploration stage
  Arms: Extended Phase Dose Group

SUMMARY:
This trial adopts an open, randomized, parallel controlled, multicenter clinical trial design planning to enroll patients with polycythemia vera who are resistant/intolerant to hydroxyurea or interferon。The study divided into two stages: dose exploration stage: three dose groups are tentatively set, with three subjects in each group, totaling nine subjects in each group; Dose extension stage: Based on the safety, efficacy, and pharmacokinetic results of the comprehensive dose exploration stage, 2-3 dose groups are planned to be selected for dose extension trials.

DETAILED DESCRIPTION:
The treatment goal of polycythemia vera is to avoid initial or recurrent thrombosis, control disease-related symptoms, prevent post PV MF and/or acute leukemia transformation after polycythemia vera. Almost all PV patients have non receptor type Janus kinase 2 (JAK2) gene mutations, typically JAK2 V617F. This drug is intended for patients with myeloproliferative neoplasms (MPN), mainly including moderate to high-risk myelofibrosis (FM) (including primary myelofibrosis (PMF)), post polycythemia vera myelofibrosis (PPV-MF), and post thrombocytopenia myelofibrosis (PET-MF), polycythemia vera (PV), and primary thrombocytosis (ET).

Flonoltinib Maleate (FM), a triple target inhibitor of JAK2/FLT3/CDK6, has the potential to inhibit JAK2 signaling pathway activity and treat bone marrow proliferative tumors.

This trial adopts an open, randomized, parallel controlled, multicenter clinical trial design. The plan is to recruit patients with polycythemia vera who are resistant/intolerant to hydroxyurea or interferon. The study is divided into two stages: dose exploration stage: three dose groups are tentatively set, with three subjects in each group,for a total of 9 subjects; Dose extension phase: Based on the safety, efficacy, and pharmacokinetic results of the comprehensive dose exploration phase, it is planned to select 2-3 dose groups for dose extension trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years old and gender not limited when signing the informed consent form;
2. Diagnosed as PV according to WHO standards (2016 edition), and resistant/intolerant to hydroxyurea or interferon treatment (refer to attachments 1 and 2);
3. When screening, the peripheral blood primitive cells are 0%;
4. Meet any of the following criteria and achieve HCT<= 45% before randomization/enrollment:

1)At least 2 venous bloodletting and/or apheresis treatments have been performed within 24 weeks prior to screening, with a minimum interval of 4 weeks between each treatment, and at least 1 treatment has occurred within 16 weeks prior to screening; 2)At least one venous bloodletting and/or apheresis treatment has been performed within the 16 weeks and HCT>45% at the time of screening; 5.When screening, laboratory test indicators meet the following criteria: neutrophil count >= 1.0 × 10 ^ 9/L, platelet count >= 100 × 10 ^ 9/L and <= 1000 × 10 ^ 9/L; ALT and AST<= 2.5 × ULN; TBIL<=2.0×ULN; Serum creatinine <= 1.5 × ULN; 6.ECOG 0-2 points; 7.Can understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Individuals with allergies or suspected allergies to the test drug and its excipients;
2. The toxic reactions of previous anti-cancer treatments have not recovered to grade 1 or below (excluding hair loss, blood routine and blood biochemical indicators refer to inclusion criteria 4 and 5), or have not fully recovered from previous surgeries (having undergone major surgery within 4 weeks);
3. In addition to PV, any other myeloproliferative neoplasms (MPN), including post polycythemia vera myelofibrosis (PPV-MF), may also be present;
4. Any active infections that require systemic treatment (oral, intravenous, subcutaneous, intramuscular, etc.) during screening;
5. Patients with swallowing difficulties, chronic diarrhea, or oral absorption disorders are included in the screening process;
6. Patients with basic diseases that are difficult to control in combination with drug treatment during screening, including but not limited to: diabetes, hypertension , peripheral neuropathy ;
7. Screening for individuals who have experienced congestive heart failure (NYHA class III or above), unstable angina, myocardial infarction, cerebrovascular accidents with functional impairment, or require treatment for arrhythmia within the past 6 months;
8. Individuals with QTcF>450 ms (male) and QTcF>470 ms (female) on electrocardiogram during screening;
9. Individuals who have experienced active tuberculosis infection within the past year prior to screening, or those whose tuberculosis related test results indicate latent infection during screening;
10. Patients who have undergone splenectomy or splenic radiotherapy in the past;
11. When screening, any of the following situations exist: a) Hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) is positive, and HBV-DNA detection is positive or above the upper limit of normal value; b) HCV antibody positive and HCV-RNA detection positive; c) Positive for anti Treponema pallidum antibody (TP Ab) and positive for Treponema pallidum non-specific antibody (PRP or TRUST) detection; d) Positive for Human Immunodeficiency Virus Antibody (HIV Ab);
12. Individuals with epilepsy or mental illnesses requiring medication during screening (excluding insomnia);
13. Individuals who have suffered from other malignant tumors within the past 5 years prior to the first administration (excluding cured carcinoma in situ and basal cell carcinoma of the skin);
14. Patients with congenital or acquired bleeding disorders or active thrombotic disorders during screening;
15. Combining other serious diseases during screening may affect patient safety or compliance, according to researchers;
16. Within 2 weeks prior to trial administration or within 5 half lives (whichever is longer), any therapeutic PV drugs have been used, including hydroxyurea, recombinant interferon - α (long-acting recombinant interferon - α treatment needs to be discontinued for 4 weeks), JAK inhibitors (such as Ruxolitinib), 32P (needs to be discontinued for 8 weeks), Busulfan, etc;
17. Patients who receive treatment with other clinical trial drugs or clinical trial medical devices before screening and have not fully eluted for at least 5 half lives or 1 month (whichever is longer);
18. Pregnant or lactating women;
19. Individuals who have the ability to conceive but refuse to use contraceptive measures during the trial period ;and within 6 months after the trial ends;
20. Vaccination with active or attenuated vaccines within 4 weeks prior to screening;
21. Researchers believe that there are other factors that are not suitable for participating in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved HCT control | At the end of the 28th week
  Achieve HCT<45% without undergoing venous bloodletting or apheresis treatmen

SECONDARY OUTCOMES:
The proportion of subjects who achieved complete hematological remission | week 28 and 52
  Without undergoing venous bloodletting or apheresis, achieve HCT<45%, PLT <= 400×10^9/L, and WBC<10×10^9/L
The duration of HCT control | The time elapsed from the date when HCT control was first recorded from the start of Day 29 treatment to the date when HCT increased to >= 45%
  The duration of HCT control (defined as the time elapsed from the date when HCT control was first recorded from the start of Day 29 treatment to the date when HCT increased to >= 45%)
Changes in the total symptom score of MPN-SAF TSS scale | week 16, 28, 40, and 52
  The MPN-SAF-TSS is used to assess the symptom burden of patients with myeloproliferative neoplasms. The questionnaire also reflects the quality of life of patients to a certain extent. During the diagnosis and treatment process, the MPN-10 questionnaire includes 10 sub symptoms (fatigue, early satiety, abdominal discomfort, poor activity, lack of concentration, night sweats, skin itching, bone pain, fever, and weight loss). Each item is graded from 0 (none) to 10 (heaviest), with a total score of 0-100 points. The higher the total score, the heavier the symptom burden.
Proportion of subjects who did not experience thrombosis or bleeding events | week 28 and 52
  Proportion of subjects who did not experience thrombosis or bleeding events at the end of treatment in weeks 28 and 52
Changes in gene mutation burden relative to baseline | week 28 and 52
  Subjects with JAK2V617F quantification>0% during the screening period will undergo JAK2V617F quantification testing at weeks 28 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences (IHCAMS); Ting Niu, Doctor, Principal Investigator — West China Hospital; Wei Yang, Doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences (IHCAMS), Tianjin, China

IPD SHARING:
Plan to Share IPD: No